CLINICAL TRIAL: NCT04278261
Title: A Prospective, Single-center, Randomized Controlled Trial Comparing the Functional and Oncological Outcomes of High-frequency Irreversible Electroporation and Laparoscopic Radical Prostatectomy in Men With Localized Prostate Cancer
Brief Title: Comparison H-FIRE and Laparoscopic RP in Treating Men With Localized Prostate Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HIRE-FR-2019001
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Prostate Cancer; Treatment
Keywords: Focal therapy; Radical prostatectomy; high-frequency Irreversible electroporation; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Focal therapy (Experimental): Using focal therapy(high-frequency Irreversible electroporation) to treat patients with localized Prostate cancer
  Interventions: Procedure: Focal therapy(high-frequency irreversible electroporation)
- Radical prostatectomy (Active Comparator): Using laparoscopic radical prostatectomy to treat patients with localized Prostate cancer
  Interventions: Procedure: laparoscopic radical prostatectomy

INTERVENTIONS:
Procedure: Focal therapy(high-frequency irreversible electroporation) — High-frequency irreversible electroporation will be performed via the perineum with the guidance of ultrasound under general anaesthesia to the patient with localized prostate cancer
  Arms: Focal therapy
Procedure: laparoscopic radical prostatectomy — Laparoscopic radical prostatectomy
  Arms: Radical prostatectomy

SUMMARY:
This trial is comparing the functional and oncological outcomes in treating men with prostate cancer between high-frequency irreversible electroporation and laparoscopic radical prostatectomy.

DETAILED DESCRIPTION:
Two hundred and sixteen patients with localized prostate cancer will include in this study. The clinical trial validation process will be as follows: (1) all patients are randomly divided into two arms: arm 1, high-frequency irreversible electroporation; group 2, laparoscopic radical prostatectomy. The primary outcome is the urinary function and sexual function.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than 80 years old.
2. PSA<20ng/ml.
3. Clinical stage ≤T2c.
4. Biopsy Gleason score ≤4+4.
5. No evidence of metastasis.
6. Fully understand the clinical trial protocol and sign the informed consent

Exclusion Criteria:

1. Any previous treatment to PCa.
2. Any previous surgery within 3 months.
3. Contraindications to MRI, bone scan, or PSMA-PET (eg, metal implant, contrast agent allergy).
4. History of any other malignant tumour.
5. Any other conditions that make the investigator judge that participants are not suitable for this trial.

Max Age: 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
urinary function measured by ICIQ | 4 weeks
  The urinary function will be measured by ICIQ (International Consultation on Incontinence Questionnaire) score
urinary function measured by ICIQ | 6 weeks
  The urinary function will be measured by ICIQ (International Consultation on Incontinence Questionnaire) score
urinary function measured by ICIQ | 12 weeks
  The urinary function will be measured by ICIQ (International Consultation on Incontinence Questionnaire) score
urinary function measured by ICIQ | 6 months
  The urinary function will be measured by ICIQ (International Consultation on Incontinence Questionnaire) score
urinary function measured by ICIQ | 12 months
  The urinary function will be measured by ICIQ (International Consultation on Incontinence Questionnaire) score
urinary function measured by ICIQ | 24 months
  The urinary function will be measured by ICIQ (International Consultation on Incontinence Questionnaire) score
urinary function measured by EPIC | 4 weeks
  The urinary function will be measured by EPIC (Expanded Prostate Cancer Index Composite) urinary domain function score
urinary function measured by EPIC | 6 weeks
  The urinary function will be measured by EPIC (Expanded Prostate Cancer Index Composite) urinary domain function score
urinary function measured by EPIC | 12 weeks
  The urinary function will be measured by EPIC (Expanded Prostate Cancer Index Composite) urinary domain function score
urinary function measured by EPIC | 6 months
  The urinary function will be measured by EPIC (Expanded Prostate Cancer Index Composite) urinary domain function score
urinary function measured by EPIC | 12 months
  The urinary function will be measured by EPIC (Expanded Prostate Cancer Index Composite) urinary domain function score
urinary function measured by EPIC | 24 months
  The urinary function will be measured by EPIC (Expanded Prostate Cancer Index Composite) urinary domain function score
urinary function measured by separate EPIC pad-use item | 4 weeks
  The urinary function will be measured by a separate EPIC pad-use item
urinary function measured by separate EPIC pad-use item | 6 weeks
  The urinary function will be measured by a separate EPIC pad-use item
urinary function measured by separate EPIC pad-use item | 12 weeks
  The urinary function will be measured by a separate EPIC pad-use item
urinary function measured by separate EPIC pad-use item | 6 months
  The urinary function will be measured by a separate EPIC pad-use item
urinary function measured by separate EPIC pad-use item | 12 months
  The urinary function will be measured by a separate EPIC pad-use item
urinary function measured by separate EPIC pad-use item | 24 months
  The urinary function will be measured by a separate EPIC pad-use item
urinary function measured by IPSS | 4 weeks
  The urinary function will be measured by IPSS (International Prostate Symptom Score)
urinary function measured by IPSS | 6 weeks
  The urinary function will be measured by IPSS (International Prostate Symptom Score)
urinary function measured by IPSS | 12 weeks
  The urinary function will be measured by IPSS (International Prostate Symptom Score)
urinary function measured by IPSS | 6 months
  The urinary function will be measured by IPSS (International Prostate Symptom Score)
urinary function measured by IPSS | 12 months
  The urinary function will be measured by IPSS (International Prostate Symptom Score)
urinary function measured by IPSS | 24 months
  The urinary function will be measured by IPSS (International Prostate Symptom Score)
sexual function measured by EPIC | 4 weeks
  The sexual function will be measured by EPIC (Expanded Prostate Cancer Index Composite) sexual function score
sexual function measured by EPIC | 6 weeks
  The sexual function will be measured by EPIC (Expanded Prostate Cancer Index Composite) sexual function score
sexual function measured by EPIC | 12 weeks
  The sexual function will be measured by EPIC (Expanded Prostate Cancer Index Composite) sexual function score
sexual function measured by EPIC | 6 months
  The sexual function will be measured by EPIC (Expanded Prostate Cancer Index Composite) sexual function score
sexual function measured by EPIC | 12 months
  The sexual function will be measured by EPIC (Expanded Prostate Cancer Index Composite) sexual function score
sexual function measured by EPIC | 24 months
  The sexual function will be measured by EPIC (Expanded Prostate Cancer Index Composite) sexual function score
sexual function measured by IIEF-5 | 4 weeks
  The sexual function will be measured by IIEF-5 (5-item version of the International Index of Erectile Function)
sexual function measured by IIEF-5 | 6 weeks
  The sexual function will be measured by IIEF-5 (5-item version of the International Index of Erectile Function)
sexual function measured by IIEF-5 | 12 weeks
  The sexual function will be measured by IIEF-5 (5-item version of the International Index of Erectile Function)
sexual function measured by IIEF-5 | 6 months
  The sexual function will be measured by IIEF-5 (5-item version of the International Index of Erectile Function)
sexual function measured by IIEF-5 | 12 months
  The sexual function will be measured by IIEF-5 (5-item version of the International Index of Erectile Function)
sexual function measured by IIEF-5 | 24 months
  The sexual function will be measured by IIEF-5 (5-item version of the International Index of Erectile Function)

SECONDARY OUTCOMES:
Number of patients with Disease progression | 24 months
  is defined either of the following items: (1) clinical evidence of progression (any of the positive results from the bone scan, pelvic MRI/CT, PSMA-PET MR/CT); (2) a positive biopsy (for the H-FIRE arm only); (3) biochemical failure (BCR, for the RP arm only, defined as a serum PSA level higher than 0.4 ng/ml after surgery)
Bowel function | 4 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel function score
Bowel function | 6 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel function score
Bowel function | 12 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel function score
Bowel function | 6 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel function score
Bowel function | 12 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel function score
Bowel function | 24 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel function score
Quality of life measure by EORTC QLQ-C30 | 4 weeks
  measured by EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 module)
Quality of life measure by EORTC QLQ-C30 | 6 weeks
  measured by EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 module)
Quality of life measure by EORTC QLQ-C30 | 12 weeks
  measured by EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 module)
Quality of life measure by EORTC QLQ-C30 | 6 months
  measured by EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 module)
Quality of life measure by EORTC QLQ-C30 | 12 months
  measured by EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 module)
Quality of life measure by EORTC QLQ-C30 | 24 months
  measured by EORTC QLQ-C30 (European Organization for Research and Treatment of Cancer Quality-of-Life Questionnaire-Core 30 module)
Quality of life measure by EPIC urinary domain bother score | 4 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) urinary domain bother score
Quality of life measure by EPIC urinary domain bother score | 6 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) urinary domain bother score
Quality of life measure by EPIC urinary domain bother score | 12 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) urinary domain bother score
Quality of life measure by EPIC urinary domain bother score | 6 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) urinary domain bother score
Quality of life measure by EPIC urinary domain bother score | 12 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) urinary domain bother score
Quality of life measure by EPIC urinary domain bother score | 24 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) urinary domain bother score
Quality of life measure by EPIC sexual domain bother score | 4 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) sexual domain bother score
Quality of life measure by EPIC sexual domain bother score | 6 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) sexual domain bother score
Quality of life measure by EPIC sexual domain bother score | 12 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) sexual domain bother score
Quality of life measure by EPIC sexual domain bother score | 6 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) sexual domain bother score
Quality of life measure by EPIC sexual domain bother score | 12 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) sexual domain bother score
Quality of life measure by EPIC sexual domain bother score | 24 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) sexual domain bother score
Quality of life measure by EPIC bowel domain bother score | 4 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel domain bother score
Quality of life measure by EPIC bowel domain bother score | 6 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel domain bother score
Quality of life measure by EPIC bowel domain bother score | 12 weeks
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel domain bother score
Quality of life measure by EPIC bowel domain bother score | 6 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel domain bother score
Quality of life measure by EPIC bowel domain bother score | 12 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel domain bother score
Quality of life measure by EPIC bowel domain bother score | 24 months
  measured by EPIC(Expanded Prostate Cancer Index Composite) bowel domain bother score
Quality of life measure by HADS | 4 weeks
  measured by Hospital Anxiety and Depression Scale (HADS)
Quality of life measure by HADS | 6 weeks
  measured by Hospital Anxiety and Depression Scale (HADS)
Quality of life measure by HADS | 12 weeks
  measured by Hospital Anxiety and Depression Scale (HADS)
Quality of life measure by HADS | 6 months
  measured by Hospital Anxiety and Depression Scale (HADS)
Quality of life measure by HADS | 12 months
  measured by Hospital Anxiety and Depression Scale (HADS)
Quality of life measure by HADS | 24 months
  measured by Hospital Anxiety and Depression Scale (HADS)
Rates of primary treatment failure | 24 months
  defined as biopsy show cancer remain at 6 months after H-FIRE procedure, or a PSA level 0.4ng/ml or higher at 3 months after RP procedure
Rates of adjuvant therapy | 4 weeks
  defined as need the adjuvant therapy including androgen-deprivation therapy, radiotherapy, chemotherapy, and salvage surgery
Rates of adjuvant therapy | 6 weeks
  defined as need the adjuvant therapy including androgen-deprivation therapy, radiotherapy, chemotherapy, and salvage surgery
Rates of adjuvant therapy | 12 weeks
  defined as need the adjuvant therapy including androgen-deprivation therapy, radiotherapy, chemotherapy, and salvage surgery
Rates of adjuvant therapy | 6 months
  defined as need the adjuvant therapy including androgen-deprivation therapy, radiotherapy, chemotherapy, and salvage surgery
Rates of adjuvant therapy | 12 months
  defined as need the adjuvant therapy including androgen-deprivation therapy, radiotherapy, chemotherapy, and salvage surgery
Rates of adjuvant therapy | 24 months
  defined as need the adjuvant therapy including androgen-deprivation therapy, radiotherapy, chemotherapy, and salvage surgery
Perioperative data (operative time) | 1 month
  operative time
Perioperative data (hemoglobin loss) | 1 month
  hemoglobin loss
Perioperative data (blood transfusion) | 1 month
  the number of patients need blood transfusion
Perioperative data (the length of hospital stay) | 1 month
  the length of hospital stay
Perioperative data(the length of indwelling catheter stay) | 1 month
  the length of indwelling catheter stay
Pain (measured by a surgical pain scale range from 0 to 10) | 24 hours
  measured by a surgical pain scale range from 0 to 10
Pain (measured by a surgical pain scale range from 0 to 10) | 2 weeks
  measured by a surgical pain scale range from 0 to 10
Pain (measured by a surgical pain scale range from 0 to 10) | 4 weeks
  measured by a surgical pain scale range from 0 to 10
Pain (measured by a surgical pain scale range from 0 to 10) | 6 weeks
  measured by a surgical pain scale range from 0 to 10
Pain (measured by a surgical pain scale range from 0 to 10) | 12 weeks
  measured by a surgical pain scale range from 0 to 10
Pain (measured by a surgical pain scale range from 0 to 10) | 6 months
  measured by a surgical pain scale range from 0 to 10
Adverse effect | 24 months
  identified by the Common Terminology Criteria for Adverse Events (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Wang, MD, Principal Investigator — Shanghai East Hospital,Tongji University School of Medicine
Locations (1):
- Shanghai East Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No